CLINICAL TRIAL: NCT03335384
Title: The Relationship Between Pulmonary Function Measures and Transdiaphragmatic Measures in Duchenne Muscular Dystrophy Subjects
Brief Title: Relationship Between PFTs and Pdi in DMD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not approved
Sponsor: University of Minnesota (Other)
Collaborators: Fairview Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001062
Record Dates: First submitted 2017-10-12; First posted 2017-11-07 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Cross-sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Measurement of Pdi (Experimental): Two small balloons, which are attached to small, flexible tubes, will be put into the esophagus (food tube) and stomach through the nose. Each balloon is about 2 inches long (deflated) and about the width of a pencil tip. A gastric balloon will be inserted into subject's stomach while an esophageal balloon will be inserted into the subject's esophagus. To reduce any discomfort with this procedure, lidocaine gel or spray will be put into the subject's nose and administered to the back of the throat before the balloon. In addition, swallowing water during the procedure will help to reduce any gagging sensation and will assure that the balloon goes into the esophagus.
  Interventions: Diagnostic Test: Esophageal Balloon; Diagnostic Test: Gastric Balloon
- Measurement of SNIPs (Experimental): While the gastric and esophageal balloon catheters are in place, the subject will be asked to perform a maximal sniff maneuver (SNIP) while one nostril is occluded with a plug containing a nasal pressure transducer to measure airway pressure during maximal inspiration. The distal end of the pressure catheter will be connected to a hand held pressure meter to display peak pressure and to provide you visual feedback. This maneuver will be performed 10 times.
  Interventions: Diagnostic Test: Nasal Pressure Transducer

INTERVENTIONS:
Diagnostic Test: Esophageal Balloon — Small flexible catheter with deflated balloon at distal end to be inserted into the esophagus through the nose
  Arms: Measurement of Pdi
Diagnostic Test: Gastric Balloon — Small flexible catheter with deflated balloon at distal end to be inserted into the stomach through the nose
  Arms: Measurement of Pdi
Diagnostic Test: Nasal Pressure Transducer — Pressure transducer inserted into nasal plug
  Arms: Measurement of SNIPs

SUMMARY:
A cross-sectional study to explore the relationship between clinically assessed pulmonary function test (PFT) measures and transdiaphragmatic (Pdi) measures in Duchenne muscular dystrophy (DMD) as well as to explore the relationship between sniff nasal inspiratory pressure (SNIP) and transdiaphragmatic (Pdi) measures in Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
Two small balloons, which are attached to small, flexible tubes, will be put into the esophagus and stomach through your nose. Each balloon is about 2 inches long (deflated) and about the width of a pencil tip. To reduce any discomfort with this procedure, lidocaine gel or spray will be put into the subject's nose and administered to the back of the throat before the balloon. In addition, swallowing water during the procedure will help to reduce any gagging sensation and will assure that the balloon goes into the esophagus. Proper placement of the catheters will be determined using normal tidal breathing against an occluded mouthpiece with a nose clip. Once proper placement is ensured, the catheters will remain in place during your normal PFT maneuvers. Additionally, while the gastric and esophageal balloon catheters are in place, the subject will be asked to perform a maximal sniff maneuver (SNIP) while one nostril is occluded with a plug containing a distal pressure measurement catheter to measure airway pressure. The distal end of the pressure catheter will be connected to a hand held pressure meter to display peak pressure and to provide you visual feedback. This maneuver will be performed 10 times.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Duchenne muscular dystrophy

Exclusion Criteria:

* Inability to follow verbal instructions

Ages: 6 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Pdi | 1 year
  For all subjects Pdi (transdiaphragmatic pressure measures) will be assessed with gastric and esophageal balloons

SECONDARY OUTCOMES:
Evaluation of SNIP | 1 year
  For all subjects, SNIP (sniff nasal inspiratory pressures) will be assessed with a nasal pressure transducer
Evaluation of FVC | 1 year
  For all subjects, FVC (forced vital capacity) will be assessed with spirometry
Evaluation of FEV1 | 1 year
  For all subjects, FEV1 (forced expiratory volume in 1 second) will be assessed with spirometry
Evaluation of FEFmax | 1 year
  For all subjects, FEFmax (maximal forced expiratory flow) will be assessed with spirometry
Evaluation of FEF25-75 | 1 year
  For all subjects, FEF25-75 (the average forced expiratory flow during the mid (25 - 75%) portion of the FVC) will be assessed with spirometry
Evaluation of FEF50 | 1 year
  For all subjects, FEF50 (forced expiratory flow at 50% of FVC) will be assessed with spirometry
Evaluation of MIP | 1 year
  For all subjects, MIP (maximal inspiratory pressure) will be assessed with spirometry
Evaluation of MEP | 1 year
  For all subjects, MEP (maximal expiratory pressure) will be assessed with spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Snyder, PhD, Principal Investigator — University of Minnesota